CLINICAL TRIAL: NCT00534053
Title: Impact of a Mailed Educational Reminder on Fecal Occult Blood Testing (FOBT): A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Screening
Other Study IDs: 070504
Record Dates: First submitted 2007-09-20; First posted 2007-09-24 (Estimated); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Colon Cancer
Keywords: colon cancer screening; mail reminders; fecal occult blood test; compliance
MeSH Terms: conditions — Colonic Neoplasms; Patient Compliance

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 400 patients will be given a mailed educational reminder 10 days after picking up their FOBT cards from the VA laboratory.
  Interventions: Other: Mailed Educational Reminder
- 2 (No Intervention): 400 patients will not receive a mailed educational reminder to return their FOBT cards after they have picked up the FOBT cards from the VA laboratory

INTERVENTIONS:
Other: Mailed Educational Reminder — 1 page educational reminder that reminds the patient to return their FOBT cards back to the VA laboratory. In addition, it also contains reasons why colon cancer screening is important.
  Arms: 1

SUMMARY:
The purpose of our randomized controlled trial is to determine whether mailed educational reminders would increase fecal occult blood test (FOBT) card return rates and, therefore, improve patient compliance with colonrectal cancer (CRC) screening.

We will conduct a randomized, controlled trial to evaluate the hypothesis that compliance to FOBT referrals is at least 10% greater among patients who receive mailed educational reminders on the importance of CRC screening. The study will be conducted in Veteran Affairs Medical Center and surrounding VA clinics in San Diego.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the third most common cancer in men and women in the United States with an estimated 147,000 new cases and more than 56,000 deaths each year. Early detection of colon cancer and removal of precancerous adenomatous polyps have been shown to reduce its morbidity, mortality and incidence. There are several recommended CRC screening tests, including fecal occult blood test (FOBT), flexible sigmoidoscopy, air-contrast barium enema, and colonoscopy. In the VA, FOBT is the predominant screening test for CRC, however patient compliance is low. Numerous studies have evaluated patient participation in CRC screening programs and FOBT card return rates, all of which have shown patient adherence was suboptimal. To date, there are no studies that have evaluated whether mailed educational reminders can improve FOBT compliance. The purpose of our randomized controlled trial is to determine whether mailed educational reminders would increase FOBT card return rates and, therefore, improve patient compliance with CRC screening.

ELIGIBILITY:
Inclusion Criteria:

* asymptomatic men and women age 50 years or older who received screening FOBT card kits from the laboratory

Exclusion Criteria:

* are less than 50 years of age
* are inpatients
* are not undergoing routine colon cancer screening

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 775 (Actual)
Dates: Start 2007-06 (Actual); Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Our primary outcome is FOBT card return rate | 6 months

SECONDARY OUTCOMES:
Predictors of Non-compliance to fecal occult blood testing | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Samuel B Ho, M.D., Principal Investigator — UCSD, VA San Diego
Locations (1):
- Veteran Affairs Medical Center San Diego, San Diego, California, United States

REFERENCES:
- [Background] Stokamer CL, Tenner CT, Chaudhuri J, Vazquez E, Bini EJ. Randomized controlled trial of the impact of intensive patient education on compliance with fecal occult blood testing. J Gen Intern Med. 2005 Mar;20(3):278-82. doi: 10.1111/j.1525-1497.2005.40023.x. PMID 15836533
- [Derived] Lee JK, Reis V, Liu S, Conn L, Groessl EJ, Ganiats TG, Ho SB. Improving fecal occult blood testing compliance using a mailed educational reminder. J Gen Intern Med. 2009 Nov;24(11):1192-7. doi: 10.1007/s11606-009-1087-5. Epub 2009 Sep 23. PMID 19774423